CLINICAL TRIAL: NCT01494701
Title: An Open-label, Escalating Dose Study to Assess the Safety, Tolerability and Dose-range Finding of a Single Intrathecal Dose of ISIS 396443 in Patients With Spinal Muscular Atrophy
Brief Title: An Open-label Safety, Tolerability, and Dose-range Finding Study of Nusinersen (ISIS 396443) in Participants With Spinal Muscular Atrophy (SMA)
Acronym: SMNRx
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISIS 396443 - CS1
Expanded Access: NCT02865109 (No longer available)
Record Dates: First submitted 2011-12-13; First posted 2011-12-19 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Spinal Muscular Atrophy
Keywords: Spinal Muscular Atrophy; SMA; SMN; SMNRx; ISIS-SMNRx; ISIS-SMN Rx; ISIS 396443; IONIS-SMNRx; IONIS-SMN Rx; Spinraza
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — nusinersen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (n=6) (Experimental)
  Interventions: Drug: nusinersen
- Cohort 2 (n=6) (Experimental)
  Interventions: Drug: nusinersen
- Cohort 3 (n=6) (Experimental)
  Interventions: Drug: nusinersen
- Cohort 4 (n=10) (Experimental)
  Interventions: Drug: nusinersen

INTERVENTIONS:
Drug: nusinersen — Administered by intrathecal (IT) injection
  Other Names: ISIS 396443; BIIB058; Spinraza; IONIS-SMN Rx; ISIS SMNRx

SUMMARY:
This objectives of this study are to evaluate the safety, tolerability, and pharmacokinetics of a single dose of nusinersen (ISIS 396443) administered intrathecally to participants with Spinal Muscular Atrophy (SMA).

DETAILED DESCRIPTION:
This study was conducted and the protocol was registered by Ionis Pharmaceuticals, Inc.

In August 2016, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Key Inclusion Criteria:

* Documented Survival Motor Neuron1 (SMN1) homozygous gene deletion
* Clinical signs attributable to Spinal Muscular Atrophy (SMA)
* Able to complete all study procedures, measurements and visits and parent/participant has adequately supportive psychosocial circumstances, in the opinion of the investigator
* Estimated life expectancy > 2 years from Screening
* Meets age-appropriate institutional criteria for use of anesthesia/sedation, if use is planned for study procedure

Key Exclusion Criteria:

* Respiratory insufficiency defined by the need for invasive or non-invasive ventilation during a 24 hour period
* Presence of a gastric feeding tube
* Previous scoliosis surgery or scoliosis surgery planned during the duration of the study that would interfere with the lumbar puncture (LP) injection procedure
* Hospitalization for surgery or pulmonary event within the last 2 months or planned during the study
* Presence of an untreated or inadequately treated active infection requiring systemic antiviral or antimicrobial therapy
* History of brain or spinal cord disease that would interfere with LP procedures or cerebrospinal fluid (CSF) circulation
* Presence of an implanted shunt for the draining of CSF or an implanted Central Nervous System (CNS) catheter
* History of bacterial meningitis
* Clinically significant abnormalities in hematology or clinical chemistry parameters
* Treatment with another investigational drug, biological agent, or device within 1-month of Screening or 5 half-lives of study agent whichever is longer. Any history of gene therapy or cell transplantation
* Ongoing medical condition that would interfere with the conduct and assessments of the study. Examples are medical disability (e.g. wasting or cachexia, severe anemia, etc.) that would interfere with the assessment of safety or would compromised the ability of the participant to undergo study procedures

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2011-11-30 (Actual); Primary Completion 2013-01-31 (Actual); Study Completion 2013-01-31 (Actual)

PRIMARY OUTCOMES:
Number of participants that experience Adverse Events (AEs) and Serious Adverse Events | Up to 88 Days
Number of participants with clinically significant neurological examination abnormalities | Up to 88 Days
Number of participants with clinically significant vital sign abnormalities | Up to 88 Days
Number of participants with clinically significant physical examination abnormalities | Up to 88 Days
Number of participants with clinically significant weight abnormalities | Up to 88 Days
Number of participants with clinically significant laboratory parameters | Up to 88 Days
Number or participants with clinically significant cerbrospinal fluid (CSF) laboratory parameters | Up to 88 Days
Number of participants with clinically significant electrocardiograms (ECGs) abnormalities | Up to 88 Days
Number of participants who use concomitant medications | Up to 88 Days
PK parameters of nusinersen (ISIS 396443): Maximum observed plasma drug concentration (Cmax) | Plasma at 1, 2, 4 and 20 hours after dosing
PK parameters of nusinersen: Time to reach maximum observed concentration (Tmax) | Plasma at 1, 2, 4 and 20 hours after dosing
PK parameters of nusinersen: Area under the plasma concentrations time curve from the time of the intrathecal (IT) dose to the last collected sample (AUCinf) | Plasma at 1, 2, 4 and 20 hours after dosing
PK parameters of nusinersen (ISIS 396443): Apparent terminal elimination half-life (t1/2), if possible | Plasma at 1, 2, 4 and 20 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (4):
- United States (4):
  - Children's Hospital Boston, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - UT Southwestern Medical Center - Children's Medical Center Dallas, Dallas, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah

REFERENCES:
- [Derived] Darras BT, Farrar MA, Mercuri E, Finkel RS, Foster R, Hughes SG, Bhan I, Farwell W, Gheuens S. An Integrated Safety Analysis of Infants and Children with Symptomatic Spinal Muscular Atrophy (SMA) Treated with Nusinersen in Seven Clinical Trials. CNS Drugs. 2019 Sep;33(9):919-932. doi: 10.1007/s40263-019-00656-w. PMID 31420846
- [Derived] Hache M, Swoboda KJ, Sethna N, Farrow-Gillespie A, Khandji A, Xia S, Bishop KM. Intrathecal Injections in Children With Spinal Muscular Atrophy: Nusinersen Clinical Trial Experience. J Child Neurol. 2016 Jun;31(7):899-906. doi: 10.1177/0883073815627882. Epub 2016 Jan 27. PMID 26823478
- See also: Cure SMA — http://www.curesma.org
- See also: Muscular Dystrophy Association — http://mda.org/disease/spinal-muscular-atrophy
- See also: National Organization for Rare Diseases — http://www.rarediseases.org
- See also: Clinical Study Report (CSR) Synopsis - a results summary — http://clinicalresearch.biogen.com/Content/Studies/CS1%20Biogen.com%20Packet.pdf